CLINICAL TRIAL: NCT07297212
Title: A Phase II, Multi-site, Open-label Trial Evaluating the Safety and Efficacy of BNT327 and Bevacizumab as Monotherapy and BNT327 in Combination With Temozolomide in Patients With Recurrent Glioblastoma
Brief Title: A Clinical Trial Testing the Safety of BNT327 (an Investigational Drug) and How Well it Works in Patients With Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Bristol-Myers Squibb (Industry); BioNTech (Shanghai) Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-10
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Glioblastoma
Keywords: Bispecific antibody; Immunotherapy; Immunotherapy in combination with chemotherapy; Brain tumor; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor(-A) (VEGF-A)
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Pumitamig Monotherapy (Experimental)
  Interventions: Drug: Pumitamig
- Arm 2: Bevacizumab Monotherapy (Experimental)
  Interventions: Drug: Bevacizumab
- Arm 3: Pumitamig + temozolomide (Experimental)
  Interventions: Drug: Pumitamig; Drug: Temozolomide

INTERVENTIONS:
Drug: Pumitamig — Intravenous (IV) infusion
  Other Names: PM8002; BNT327; BMS-986545
  Arms: Arm 1: Pumitamig Monotherapy; Arm 3: Pumitamig + temozolomide
Drug: Bevacizumab — IV infusion
  Arms: Arm 2: Bevacizumab Monotherapy
Drug: Temozolomide — Oral
  Arms: Arm 3: Pumitamig + temozolomide

SUMMARY:
This multi-site Phase II study will enroll adults with histologically confirmed diagnosis of World Health Organization (WHO) Grade IV glioblastoma (GBM) consistent with WHO central nervous system (CNS) 2021 criteria who have received prior first-line treatment including with at least radiotherapy and temozolomide, with a Karnofsky performance status (KPS) ≥60, adequate organ function, and at least one measurable lesion according to the response assessment in neuro-oncology (RANO) 2.0 criteria.

DETAILED DESCRIPTION:
Participants will be randomized to the two treatment Arms 1 and 2. After sponsor evaluation of the initial safety and efficacy signals from Arm 1, it will be determined whether to initiate Arm 3. There will be a screening period of up to 28 days, followed by a treatment period lasting up to 2 years. Participants will be followed-up for safety for up to 90 days after the last dose of study treatment or until the participant initiates new anticancer treatment (e.g., systemic, radiotherapy/surgery). Thereafter, survival follow-up will be conducted until the participant dies, the participant withdraws consent for survival status follow-up, loss of contact, or study termination (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-75 years of age at the time of giving informed consent. Local laws will be followed if the age at consent is older.
* Have a histologically confirmed diagnosis of WHO Grade IV GBM consistent with WHO CNS 2021 criteria.
* Have recurrent supratentorial GBM who have received prior first-line treatment with at least radiotherapy and temozolomide.
* Have first recurrence documented by magnetic resonance imaging (MRI), with an interval of at least 12 weeks after the end of prior radiotherapy unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field.
* Have been clinically evaluated as having relapsed or progressed disease with at least one measurable lesion as the targeted lesion based on RANO 2.0 criteria.
* Have KPS ≥60.
* Can swallow the medication and maintain oral administration.
* Have a baseline brain MRI, not more than 14 days before starting the study treatment.
* Have a stable dose of steroids ≥7 days before the contrast-enhanced scan.
* Have adequate organ function, as defined in the protocol.

Exclusion Criteria:

* Have received any of the following therapies or drugs before study enrollment:

  * Any anticancer therapies, including systemic, palliative, biologic, immunostimulatory, or immunosuppressive treatment within 4 weeks (or five half-lives, whichever is longer) before starting the study treatment.
  * PD(L)-1/VEGF bispecific antibodies, anti-VEGF drugs, cluster of differentiation (CD)137 agonists or other immune checkpoint blockade therapies including monotherapy with either category or combinations thereof.
  * Systemic corticosteroids (at a dosage greater than 2 mg/day of dexamethasone or an equivalent dose of other corticosteroids) within 7 days before starting the study treatment.
  * Vaccinations with live attenuated vaccine(s) within 4 weeks before starting the study treatment.
  * Broad-spectrum intravenous antibiotics therapy within 2 weeks before starting the study treatment.
  * Any non-study investigational medicinal product within five half-lives of the first dose or within 4 weeks, whichever is longer, before starting the study treatment in this study or ongoing participation in the active treatment phase of another interventional clinical study.
  * Antiplatelet drugs, such as aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine or cilostazol, etc., within 10 days before starting the study treatment to avoid inclusion of participants who have used platelet aggregation inhibitors before the study.
* Have had more than one recurrence of GBM.
* Are allergic to dacarbazine and temozolomide.
* Have known leptomeningeal disease, gliomatosis cerebri, extracranial disease, or multicentric disease.
* Have been diagnosed with secondary GBM (i.e., glioblastomas that progress from low grade diffuse astrocytoma or anaplastic astrocytoma).
* Have previously received radiotherapy with anything other than standard radiotherapy (i.e., focally directed radiation).
* Have received prior interstitial brachytherapy, interstitial thermal therapy, implanted chemotherapy, or therapeutics delivered by local injection or convection-enhanced drug delivery. Participants who had prior treatment with Gliadel® wafers and who had concurrent use of devices such as Tumor Treating Fields are excluded.
* Have uncontrolled hypertension or poorly controlled diabetic conditions as specified in the protocol before study enrollment.
* Are unable (due to existent medical condition, e.g., pacemaker or implantable cardioverter defibrillator device) or unwilling to have a head contrast-enhanced MRI.
* Have undergone major surgery, open biopsy, or significant traumatic injury within 28 days before starting the study treatment, or a planned/anticipated need for major surgery during the study treatment period. Placement of vascular infusion devices is allowed. Note: If participant has had major surgery, they must have recovered adequately from the toxicity and/or complications from the treatment prior to the initiation of study treatment.
* Have received allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Have had other malignant tumors within 5 years before starting the study treatment. Exception: those who have been cured with local treatment (such as basal cell or squamous-cell carcinoma of the skin, superficial or noninvasive bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary carcinoma of thyroid and early-stage prostate cancer).
* Have any of the following heart conditions within 6 months before starting the study treatment:

  * Myocardial infarction, unstable angina, acute coronary syndrome, coronary artery bypass grafting, congestive heart failure, aortic dissection, stroke, cerebrovascular accident or other Grade 3 and above cardiovascular events.
  * New York Heart Association functional classification ≥II heart failure or left ventricular ejection fraction <50%.
  * Ventricular arrhythmias requiring clinical intervention, second- to third-degree atrioventricular block, or congenital long QT syndrome. Participants with stable treated cardiac arrythmia/atrial fibrillation are allowed.
  * Mean QTcF >480 ms (the electrocardiogram can be repeated at the discretion of the investigator).
  * Cardiac troponin I or T >2 × upper limit normal.
* Have serious or non-healing wounds, ulcers, or (incompletely healed) bone fracture. This includes history (within 6 months before starting the study treatment) or risk of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess or esophageal and gastric varices, or acute gastrointestinal bleeding. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Have significant risk of hemorrhage (in the opinion of the investigator) or evidence of major coagulation disorders.
* Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). However, participants who are clinically stable following treatment for these conditions (including therapeutic thoracentesis or paracentesis or with indwelling catheters, e.g., PleurX) are allowed.
* Active colitis, including infectious, radioactive, ischemic enteritis, within 4 weeks before starting the study treatment.
* Have a history of serious Grade 3 or higher immune-related adverse events that led to treatment discontinuation of a prior immunotherapy.
* History of serious allergic diseases, history of serious allergy to drugs (including unlisted investigational drug) or known allergy or intolerance to any ingredient of the study treatment
* Uncontrolled seizures after best medical therapy or other neurological conditions including clinically significant autoimmune neurological disorders which can increase risk for adverse effects or confound assessment of study outcomes as determined by the investigator.
* Have superior vena cava syndrome or symptoms of spinal cord compression.
* Have active, or a history of, pneumonitis requiring treatment with steroids, or have active or a history of interstitial lung disease.
* Have a known history of tuberculosis that was not successfully treated.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall response rate (ORR) | Up to 24 months
  For Treatment Arms 1 and 2 only. Defined as the percentage of study participants in whom a confirmed complete response (CR) or confirmed partial response (PR) (assessed by the blinded independent central review [BICR] per RANO) is observed as best overall response.
Occurrence of treatment emergent adverse events (TEAEs) by severity | From the first dose of study treatment until 90 days after the last dose of study treatment (up to 27 months)
  According to (United States National Cancer Institute) Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v5.0]). By relationship. For Treatment Arms 1 and 3 only.
Occurrence of dose interruptions, reductions or discontinuations of study treatment due to TEAEs | Up to 24 months
  For Treatment Arms 1 and 3 only.

SECONDARY OUTCOMES:
Confirmed ORR | Up to 24 months
  Defined as the percentage of study participants in whom a confirmed CR or confirmed PR (assessed by BICR and the investigator per [immunotherapy] iRANO and only per RANO 2.0 by the investigator) is observed as best overall response (for Treatment Arms 1 and 2 only).
  For Treatment Arm 3, assessment done only by BICR per RANO 2.0.
Progression free survival (PFS) | Up to 24 months
  For Treatment Arms 1 and 2 only. Defined as the time from randomization to first documented tumor progression (progressive disease assessed by BICR and investigator per RANO 2.0 and iRANO) or death from any cause, whichever occurs first.
PFS at 6 months | At 6 months from time of randomization
  For Treatment Arms 1 and 2 only. Assessed by BICR and investigator per RANO 2.0 and iRANO.
Duration of response | Up to 24 months
  For Treatment Arms 1 and 2 only. Defined as the time from first objective response (CR or PR as assessed by BICR and investigator per RANO 2.0 and iRANO) to first occurrence of objective tumor progression (progressive disease as assessed by BICR and investigator per RANO 2.0 and iRANO), or death from any cause, whichever occurs first.
Disease control rate | Up to 24 months
  For Treatment Arms 1 and 2 only. Defined as the percentage of study participants in whom a confirmed CR or confirmed PR or stable disease (assessed by BICR and investigator per RANO 2.0 and iRANO) is observed as best overall response.
Overall survival (OS) | Up to 42 months
  For Treatment Arms 1 and 2 only. Defined as the time from participant randomization to death from any cause and at 6 and 12 months.
OS rate | At 6 and 12 months
  For Treatment Arms 1 and 2 only.
Pharmacokinetic (PK) assessment: Maximum concentration (Cmax) derived from serum concentration of pumitamig | Up to 6 months from first dose of study treatment
  For Treatment Arms 1 and 3 only. At Cycle 1 and Cycle 6 as data permits.
PK assessment: Minimum concentration (Cmin) derived from serum concentration of pumitamig | Up to 6 months from first dose of study treatment
  For Treatment Arms 1 and 3 only. At Cycle 1 and Cycle 6 as data permits.
Incidence of detectable pumitamig anti-drug antibodies in serum | Up to 27 months
  For Treatment Arms 1 and 3 only. From before the first dose of study treatment until the last survival follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No